CLINICAL TRIAL: NCT05668455
Title: Comparison of Topical Hydrocortisone Versus Dexamethasone Treatment for Inflammatory Secretions of the Conjonctiva in Patients With Ocular Prostheses
Brief Title: Comparison of Topical Treatment for Inflammatory Secretions of the Conjonctiva (Patients With Ocular Prostheses)
Acronym: CRYSTAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agnes (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Laboratoires Thea (Industry)
Responsible Party: Sponsor-Investigator, Agnes, Clinical trials Project manager, Rennes University Hospital
Organization: Rennes University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC21_8901_CRYSTAL
Record Dates: First submitted 2022-10-03; First posted 2022-12-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ocular Inflammation; Ocular Prostheses
MeSH Terms: interventions — Hydrocortisone; Dexamethasone; Povidone

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, controlled, randomised, single-blind, cross-over clinical study with 2 treatments and an artificial tear.
  (First treatment (14 days) and Wash out (1month) / Second treatment treatment (14 days) and Wash out (1month) /Third treatment (14 days) and Wash out (1month)
Who Masked: Participant
Masking Description: re-labelling for clinical trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HYDROCORTISONE (Experimental): Topical corticosteroid : hydrocortisone
  Interventions: Drug: Hydrocortisone
- DEXAMETHASONE (Experimental): Topical corticosteroid : dexamethasone
  Interventions: Drug: Dexamethasone
- POVIDONE (Placebo Comparator): Topical : tear substitute
  Interventions: Other: Povidone

INTERVENTIONS:
Drug: Hydrocortisone — 1 drops 4 times a day
  Arms: HYDROCORTISONE
Drug: Dexamethasone — 1 drops 4 times a day
  Arms: DEXAMETHASONE
Other: Povidone — 1 drops 4 times a day
  Arms: POVIDONE

SUMMARY:
We propose to evaluate the efficacy of treatment with Hydrocortisone and Dexamethasone (in a cross-over design) in patients with ocular prostheses and significant functional discomfort.

DETAILED DESCRIPTION:
There are more than 100,000 eye prosthesis wearers in France. Half of these patients are bothered by secretions or sandy sensations, or even chronic pain. Various anti-inflammatory treatments are proposed without scientific basis.

A pilot study on a limited number of patients conducted in 2017 at the University Hospital of Rennes and published in 2019 showed the interest of Dexamethasone eye drops in these patients. However, this study was retrospective and not controlled.

We therefore wish to propose a prospective, placebo-controlled, single-blind clinical study to define the value of anti-inflammatory treatment in patients with ocular prostheses.

We propose to evaluate the efficacy of treatment with Hydrocortisone and Dexamethasone (in a cross-over design) in patients with ocular prostheses and significant functional discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older;
* Wearing a permanent prosthesis for more than 6 months; - Consultant in the ophthalmology department;
* Modified OSDI score ≥ 20 points out of 40 ;
* Affiliated with a health insurance scheme,
* For women of childbearing age: effective contraception (effective contraception includes oral contraception, intrauterine devices and other forms of contraception with a failure rate <1%, for the duration of the study and up to 1 week after the last dose administered)
* Have given free, informed and written consent.

Exclusion Criteria:

* Treatment with eye drop(s) (other than artificial tears or antiseptic) < 1 month;
* Concomitant treatment with CYP3A inhibitors including cobicistat containing drugs,
* Known contraindications to study treatments
* Dermal fat grafting or complicated cavity;
* Gougerot-Sjögren syndrome;
* Allergic conjunctivitis;
* Damaged prosthesis;
* Impossibility of carrying out the various tests required by the protocol for whatever reason (comprehension problems, motor disability);
* Pregnant or breastfeeding woman;
* Person already included in a RIPH1 research protocol with topical treatment of the cavity or systemic anti-inflammatory treatment and/or who could lead to a bias in the present study
* Person under legal protection (safeguard of justice, curatorship, guardianship) or person deprived of liberty.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Secretion Self-Rating Analog Scale score. | Before first treatment period of 14 days
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40 point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)
Secretion Self-Rating Analog Scale score. | After first treatment period of 14 days
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40-point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)
Secretion Self-Rating Analog Scale score. | At 1.5 month (1 Month Wash-out after first treatment, and before second treatment)
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40-point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)
Secretion Self-Rating Analog Scale score. | At 2 months (After second treatment period of 14 days)
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40-point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)
Secretion Self-Rating Analog Scale score. | At 3 months (1 Month Wash-out after second treatment, and before third treatment)
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40-point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)
Secretion Self-Rating Analog Scale score. | At 3.5 months (After third treatment period of 14 days)
  The overall score is analysed as the primary endpoint. Each sub-score is analysed independently in the secondary endpoints.
  This 40-point score is calculated as the sum of 4 criteria, each scored on 10 points.
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick)

SECONDARY OUTCOMES:
Bulbar conjunctival inflammation score | At inclusion visit (basal)
  Bulbar conjunctival inflammation score according to the grades of Saini et al. (Grade 1 to 3 : from normal to severe)
Bulbar conjunctival inflammation score | After first treatment period of 14 days
  Bulbar conjunctival inflammation score according to the grades of Saini et al. (Grade 1 to 3 : from normal to severe)
Bulbar conjunctival inflammation score | At 2 months (After second treatment period of 14 days)
  Bulbar conjunctival inflammation score according to the grades of Saini et al. (Grade 1 to 3 : from normal to severe)
Bulbar conjunctival inflammation score | At 3.5 months (After third treatment period of 14 days)
  Bulbar conjunctival inflammation score according to the grades of Saini et al. (Grade 1 to 3 : from normal to severe)
Tarsal conjunctival inflammation score according | At inclusion visit (basal)
  Tarsal conjunctival inflammation score according to the grades of Saini et al.(Grade 1 to 4 : from absent to more than one millimetre in diameter)
Tarsal conjunctival inflammation score according | After first treatment period of 14 days
  Tarsal conjunctival inflammation score according to the grades of Saini et al.(Grade 1 to 4 : from absent to more than one millimetre in diameter)
Tarsal conjunctival inflammation score according | At 2 months (After second treatment period of 14 days)
  Tarsal conjunctival inflammation score according to the grades of Saini et al.(Grade 1 to 4 : from absent to more than one millimetre in diameter)
Tarsal conjunctival inflammation score according | At 3.5 months (After third treatment period of 14 days)
  Tarsal conjunctival inflammation score according to the grades of Saini et al.(Grade 1 to 4 : from absent to more than one millimetre in diameter)
Secretion frequency | Before first treatment period of 14 days
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Secretion frequency | After first treatment period of 14 days
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Secretion frequency | At 1.5 month (Before second treatment period of 14 days
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Secretion frequency | At 2 months (After second treatment period of 14 days
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Secretion frequency | At 3 months (Before third treatment period of 14 days)
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Secretion frequency | At 3.5 months (After third treatment period of 14 days)
  Analog scale from 1 to 10 on the frequency of secretions (from never to all the time) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | Before first treatment period of 14 days
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | After first treatment period of 14 days
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | At 1.5 month (Before second treatment period of 14 days)
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | At 2 months (After second treatment period of 14 days
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | At 3 months (Before third treatment period of 14 days)
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Colour of secretions | At 3.5 months (After third treatment period of 14 days)
  Analog scale from 1 to 10 on the colour of secretions (from clear to yellow) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | Before first treatment period of 14 days
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | After first treatment period of 14 days
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | At 1.5 month (Before second treatment period of 14 days)
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | At 2 months (After second treatment period of 14 days
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | At 3 months (Before third treatment period of 14 days
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Amount of secretions | At 3.5 months (After third treatment period of 14 days)
  Analog scale from 1 to 10 on the quantity of secretions (from minimal to profuse) according to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | Before first treatment period of 14 days
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | After first treatment period of 14 days
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | At 1.5 month (Before second treatment period of 14 days)
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | At 2 months (After second treatment period of 14 days
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | At 3 months (Before third treatment period of 14 days)
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
Thickness/Viscosity of secretions | At 3.5 months (After third treatment period of 14 days)
  Analog scale from 1 to 10 on the viscosity of secretions (from liquid to very thick) to the secretion analysis scale (Jacobs et al.)
OSDI quality of life score adapted to prosthesis wearers | Before first treatment period of 14 days
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)
OSDI quality of life score adapted to prosthesis wearers | After first treatment period of 14 days
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)
OSDI quality of life score adapted to prosthesis wearers | At 1.5 month (Before second treatment period of 14 days)
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)
OSDI quality of life score adapted to prosthesis wearers | At 2 months (After second treatment period of 14 days
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)
OSDI quality of life score adapted to prosthesis wearers | At 3 months (Before third treatment period of 14 days)
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)
OSDI quality of life score adapted to prosthesis wearers | At 3.5 months (After third treatment period of 14 days)
  OSDI quality of life score adapted to prosthesis wearers, scored on 40 points (10 items with a maximum of 4 points per item) (Maucourant et al.)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Rennes _ Pontchaillou, Rennes, France